CLINICAL TRIAL: NCT01975922
Title: An Efficacy Trial of Milieu Teaching Language Intervention in Children With Language Disorders
Brief Title: Working on Rapid Language Development in Toddlers
Acronym: WORLD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Ann Kaiser, Professor, Vanderbilt University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 090904; R324A090181 (Other Grant/Funding Number: IES)
Record Dates: First submitted 2013-10-23; First posted 2013-11-05 (Estimated); Results first posted 2018-01-26 (Actual); Last update posted 2018-01-26 (Actual); Status verified 2017-06

CONDITIONS: Language Developmental Disorders
Keywords: language impairment; language disorder; language delay; late talkers; late talking
MeSH Terms: conditions — Language Development Disorders; Language Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Enhanced Milieu Teaching (Experimental): Parents receive 28 intervention sessions in which they learn to use language support strategies with their children.
  Children are assessed at baseline, 4 months after baseline, 10 months after baseline, and 16 months after baseline.
  Interventions: Behavioral: Enhanced Milieu Teaching
- Community Services (No Intervention): Children receive speech-language services in the community. Children are assessed at baseline, 4 months after baseline, 10 months after baseline, and 16 months after baseline.

INTERVENTIONS:
Behavioral: Enhanced Milieu Teaching — Enhanced Milieu Teaching (EMT) is a conversation-based model of early language intervention that uses child interest and initiations as opportunities to model and prompt language use in everyday contexts.
  Arms: Enhanced Milieu Teaching

SUMMARY:
The goal of the study is to examine the effects of teaching parents to use language support strategies on language skills in toddlers with language delays. We hypothesize that children whose parents who learn to use language support strategies at home will have greater language skills than those children whose parents do not learn the strategies.

DETAILED DESCRIPTION:
The goal of the proposed project is to conduct an efficacy trial to determine whether Enhanced Milieu Teaching (EMT) significantly improves language deficits in young children at high risk for persistent language delays. The target population is children ages 24 -36 months who exhibit significant co-occurring delays in productive and receptive language skills, who have cognitive skills within the range of normal development, and who do not have other identified disabilities. An empirically based and manualized language intervention, Enhanced Milieu Teaching (EMT), implemented by therapists and parents will be compared to community based "business as usual" services in a randomized experiment enrolling 120 children and their parents. Children assigned to the EMT group will receive 24, 1-hour sessions of direct intervention at home that will include teaching their parents to implement EMT procedures across activities. Children will be assessed at 4 time points (before and after intervention, at 6 months and 12 months post-intervention) allowing the description and comparison of individual language growth trajectories over a period of 18 months. In addition, we will examine the relation between language growth and emergent problems in behavior and social skill development to determine whether early language intervention can prevent these difficulties frequently associated with early language delays. Results from this study will determine the efficacy of parent-plus-therapist implemented EMT with a new population of children, provide evidence about the potential for preventing persistent language delays and secondary social effects of early language delays, and expand developmental theory linking persistent language delays to specific risk factors and behavioral outcomes. The results of this study will have specific policy implications related to early identification and the inclusion of young children with language delays as a target population for early intervention.

ELIGIBILITY:
Inclusion Criteria:

* Language delay

Exclusion Criteria:

* Hearing loss
* Language other than English as the home language
* Additional disabilities (e.g., autism, Down syndrome)

Ages: 24 Months to 42 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 97 (Actual)
Dates: Start 2009-09; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ann P Kaiser, PhD, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States

REFERENCES:
- [Derived] Roberts MY, Kaiser AP. Early intervention for toddlers with language delays: a randomized controlled trial. Pediatrics. 2015 Apr;135(4):686-93. doi: 10.1542/peds.2014-2134. Epub 2015 Mar 2. PMID 25733749

RESULTS

PARTICIPANT FLOW:
Groups:
- Enhanced Milieu Teaching: Parents receive 28 intervention sessions in which they learn to use language support strategies with their children.
  Children are assessed at baseline, 4 months after baseline, 10 months after baseline, and 16 months after baseline.
  Enhanced Milieu Teaching: Enhanced Milieu Teaching (EMT) is a conversation-based model of early language intervention that uses child interest and initiations as opportunities to model and prompt language use in everyday contexts.
Period: Overall Study
Arm/Group | Enhanced Milieu Teaching | Community Services
Started | 45 | 52
Completed | 45 | 43
Not Completed | 0 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Enhanced Milieu Teaching | Community Services | Total
Number analyzed (Participants) | 45 | 52 | 97
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 45 | 52 | 97
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: months] | 30.3 (5.0) | 30.6 (5.1) | 30.4 (5.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 10 | 18
  Male | 37 | 42 | 79
Region of Enrollment [Number; unit: participants]
  United States | 45 | 52 | 97

OUTCOME MEASURES:

1. Primary Outcome: Language Skills at 4 Months After Baseline as Measured by the Pre-school Language Scale - 4th Edition
Description: Pre-school Language Scale - 4th Edition (a norm-referenced measure of receptive and expressive language) This scale measures the child's expressive and receptive language by going through a standard protocol of items, beginning based on the child's age, requiring a Basal of 3 consecutive correct responses and a Ceiling of 6 consecutive incorrect responses.
  A higher score is considered better. A standard score of 100 is considered average for the child's age with scores ranging from 50-150.
Time Frame: 4 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Enhanced Milieu Teaching | Community Services
Number analyzed (Participants) | 45 | 43
units on a scale | 84 (13.9) | 80.2 (12)

2. Secondary Outcome: Expressive Vocabulary at 4 Months After Baseline
Description: Number of different words the child says during a 20-minute language sample.
Time Frame: 4 months
Measure: Mean (Standard Deviation); unit: Number of Different words
Arm/Group | Enhanced Milieu Teaching | Community Services
Number analyzed (Participants) | 45 | 43
Number of Different words | 54.87 (29.87) | 37.98 (29.97)

ADVERSE EVENTS:
Time Frame: 16 months
Description: Children are assessed and observed for adverse events based on involvement at baseline, 4 months after baseline, 10 months after baseline, and 16 months after baseline.
Arm/Group | Enhanced Milieu Teaching | Community Services
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/43
Other Adverse Events (participants affected / at risk) | 0/45 | 0/43

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No